CLINICAL TRIAL: NCT01325792
Title: Prospective, Multicenter, Observational Study Evaluate Single-Staged Open Complex Ventral Incisional Hernia Repair Using a Biosynthetic Material for Midline Fascial Closure Reinforcement
Brief Title: Open Complex Ventral Incisional Hernia Repair Using Biosynthetic Material for Midline Fascial Closure Reinforcement
Acronym: COBRA
Status: Completed | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: CS155
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Results first posted 2015-12-24 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Ventral Incisional Hernia
Keywords: Complex ventral incisional hernia repair; reapproximation of the rectus abdominis muscle; retrorectus or intraperitoneal placement technique; mobility for midline fascial closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GORE® BIO-A® Tissue Reinforcement: Single-staged open complex ventral incisional repair of primary or recurrent anterior abdominal wall hernia.
  Interventions: Device: GORE® BIO-A® Tissue Reinforcement

INTERVENTIONS:
Device: GORE® BIO-A® Tissue Reinforcement — Retrorectus or intraperitoneal placement of device to reinforce the midline fascial closure after single-staged open complex ventral incisional hernia repair of primary or recurrent anterior abdominal wall hernia.
  Other Names: Biosynthetic Mesh

SUMMARY:
Prospective, multicenter, observational study to evaluate performance of GORE® BIO-A® Tissue Reinforcement when used to reinforce midline fascial closure in single-staged open complex ventral incisional hernia repair.

DETAILED DESCRIPTION:
The study will evaluate the performance of the biosynthetic mesh when used to reinforce the midline fascial closure in single-staged open complex ventral incisional hernia repair. It is designed to test the null hypothesis that the two year recurrence rate associated with the device is greater than or equal to 50% vs the alternative hypothesis that the two year recurrence rate is less than 50%.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be informed about the study, and will have read; understood and signed the informed consent and authorization to use their PHI, as applicable
* Subjects willing and able to submit to postoperative follow-up evaluations including quality of life assessments up to 24 months after surgery
* Subjects of either gender that are at least the age of 18 years
* Subjects will have a Body-Mass Index (BMI) of < 40
* Subjects will be undergoing single-staged open complex ventral incisional hernia repair with the retrorectus or intraperitoneal placement technique of the GORE® BIO-A® Tissue Reinforcement
* Subjects in which intraoperatively their surgical field/wound is characterized either a Type 2 or Type 3 in Table 1 in Section 12.0
* Subjects with a hernia defect > 9 cm2 large when measured intraoperatively
* Subjects in which the required mobility for midline fascial closure without excessive tension to reapproximate the rectus abdominis muscle intraoperatively can be achieved
* Subjects in which one unit of GORE® BIO-A® Tissue Reinforcement will adequately reinforce the midline fascial closure with at least 4 cm of overlap laterally

Exclusion Criteria:

* Subjects who, in the surgeon's opinion, would have a difficult time comprehending or complying with the requirements of the study
* Subjects with a BMI > 40
* Subjects with evidence of pre-existing systemic infections
* Subjects with cirrhosis or are currently being treated with dialysis
* Subjects with a wound-healing disorder
* Subjects with autoimmune disorder requiring > 10mg of a corticosteroid per day
* Subjects who are immunocompromised such as, with HIV or transplant, or receiving chemo or radiation therapy
* Subjects with a hernia defect < 9 cm2 large when measured intraoperatively
* Subjects with a hernia defect requiring more than one unit of GORE® BIO-A® Tissue Reinforcement
* Subjects in which intraoperatively there is an inability to achieve retrorectus or intraperitoneal placement of the device
* Subjects in which a midline fascial closure without excessive tension cannot be achieved
* Subjects in which intraoperatively their surgical field/wound is characterized either a Type 1 or Type 4 in the Table 1 in Section 12
* Subjects in need of concomitant surgical procedures other than indicated in the protocol as acceptable
* Subject in which their complex ventral incisional hernia repair requires more than one operation to reduce hernia and close fascia, including serial excision procedures - requiring subsequent surgery to complete their hernia repair
* Subjects with a hernia repair requiring an emergent procedure, such as strangulated bowel
* Subjects in which intraoperatively untreated cancer was found

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: general and teaching hospitals
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2011-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rosen, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (9):
- United States (8):
  - UCSD Department of Surgery, San Diego, California
  - Indiana University, Indianapolis, Indiana
  - Washington University, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Case Medical Center, Case Western Reserve University, Case Western Reserve University, Cleveland, Ohio
  - Greenville Hospital System, Greenville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canisius-Wilhelmina Ziekenhuis, Nijmegen, The Netherlands, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 104 subjects recruited from 9 sites in the US and Netherlands between March 2011 and December 2012
Groups:
- Single-staged Open Complex Ventral Incisional Hernia Repair: GORE® BIO-A® Tissue Reinforcement to reinforce the midline fascial closure in single-staged open complex ventral incisional (primary or recurrent anterior abdominal wall) hernia repair.
Period: Overall Study
Arm/Group | Single-staged Open Complex Ventral Incisional Hernia Repair
Started | 104
Completed | 87
Not Completed | 17

BASELINE CHARACTERISTICS:
Groups:
- Single-staged Open Complex Ventral Incisional Hernia Repair: primary or recurrent anterior abdominal wall hernia
  GORE BIO-A Tissue Reinforcement: Retrorectus or intraperitoneal placement of device to reinforce the midline fascial closure
Arm/Group | Single-staged Open Complex Ventral Incisional Hernia Repair
Number analyzed (Participants) | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 42
Wound Classification [Number; unit: participants] — Intraoperatively assessed, based on the level of contamination present, or due to concomitant surgical procedures, the surgical field was managed to reduce or appropriately eliminate microbial contaminants. After devitalized tissue was removed and the appropriate bioburden reduction techniques completed, the resulting surgical field/wound was characterized and documented as applicable based on the surgical wound classification scheme as suggested by the Centers for Disease Control, US Department of Human Services, with modifications for inclusion of stomas.
  participants
    Clean-contaminated | 24
    Contaminated | 80
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Hernia Recurrence Rate
Description: Investigator confirmed hernia recurrence by physical examination
Time Frame: at about 24 months
Measure: Number (95% Confidence Interval); unit: % of subjects with recurrent hernia
Arm/Group | Single-staged Open Complex Ventral Incisional Hernia Repair
Number analyzed (Participants) | 87
% of subjects with recurrent hernia | 17.3 [11.0 to 26.8]

2. Secondary Outcome: Early and Long-term Complication Rates
Description: Surgical site abdominal wound event rate
Time Frame: after surgery (day 1) to 24 months
Measure: Number; unit: % of subjects with events
Arm/Group | Single-staged Open Complex Ventral Incisional Hernia Repair
Number analyzed (Participants) | 104
% of subjects with events | 29.8

ADVERSE EVENTS:
Arm/Group | GORE® BIO-A® Tissue Reinforcement
Serious Adverse Events (participants affected / at risk) | 3/104
Other Adverse Events (participants affected / at risk) | 25/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GORE® BIO-A® Tissue Reinforcement (N=104)
Bowel obstruction related to concomitant small bowel anastomoses during index surgery (Gastrointestinal disorders) | 1 (1) — Secondary outcome event
Anastomotic leak related to concomitant bowel resection during index surgery (Gastrointestinal disorders) | 2 (2) — Secondary outcome event
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GORE® BIO-A® Tissue Reinforcement (N=104)
Surgical site infection (Infections and infestations) | 19 (21) — Secondary outcome event
Surgical site seroma (General disorders) | 6 (6) — Secondary outcome event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proposed publications/public disclosures within 60 days prior to submission will be provided to sponsor for review by Investigator. Sponsor may make modifications to the proposals only as reasonably necessary to ensure the proper use of any references to itself, its trademarks, and trade names. Sponsor may correct inaccuracies in any technical specifications or descriptions of the biosynthetic material.